CLINICAL TRIAL: NCT06670924
Title: A Pragmatic Randomized Controlled Trial Comparing the Effects of Suturing Techniques for Vesico-urethral Anastomosis on One-year Voiding Function After Radical Prostatectomy
Brief Title: Suturing Techniques for Vesico-urethral Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kartal City Hospital (Other)
Responsible Party: Principal Investigator, Utku Can, Assistant professor of urology, Kartal City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: kartalcity_ucan_001
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer Surgery
Keywords: prostate cancer; vesicourethral anastomosis; voiding function; suture
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The investigators conducted a two-group, parallel-design, pragmatic study of 70 consecutive patients with clinically localised (pT1-pT2) PCa undergoing primary open RP by a well-experienced single surgical team at Dr Lutfi Kirdar City Hospital as a tertiary care institution .The optimal sample size for this study was calculated to be 70 patients (35 patients in each arm) by the power calculation (α = 0.05, β = 0.1, power: 90%) The subjects were randomly assigned to one of two treatment groups using a simple randomization procedure that involved computer-generated random numbers in Microsoft Excel.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Data were collected by an independent database administrator and stored in a password-protected Microsoft Excel file. The data files were not accessible to the surgical team or to residents or ancillary staff involved in postoperative care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Running suture (RS) (Active Comparator): Running suture technique for vesico-urethral anastomosis in open radical prostatectomy
  Interventions: Procedure: Running suture for vesico-urethral anastomosis in open radical prostatectomy
- Interrupted suture (IS) (Active Comparator): Interrupted suture technique for vesico-urethral anastomosis in open radical prostatectomy
  Interventions: Procedure: interrupted suture for vesico-urethral anastomosis in open radical prostatectomy

INTERVENTIONS:
Procedure: Running suture for vesico-urethral anastomosis in open radical prostatectomy — The surgical technique of the RS followed the description of Van Velthovens, was applied with slight modifications. Two 3/0 absorbable monofilament (polydioxanone) sutures were used. The first needle is started from bladder neck at 3 o'clock, and terminated in the urethra at 9 o'clock. After completion of the posterior anastomosis, a transurethral catheter is placed. The second sutures' needle is passed from the bladder at 9 o'clock and ended in the urethra at 3 o'clock. The bladder neck and urethra are merged by gentle traction of the anterior and posterior sutures at 3 and 9 o'clock.
  Arms: Running suture (RS)
Procedure: interrupted suture for vesico-urethral anastomosis in open radical prostatectomy — The technique described by Walsh for interrupted anastomotic suturing was applied with minor modifications. Six 3/0 absorbable monofilament (polydioxanone) sutures were placed at 1, 3, 5, 7, 9 and 11 o'clock to accomplish the vesicourethral anastomosis.
  Arms: Interrupted suture (IS)

SUMMARY:
Radical prostatectomy (RP) is the most common curative treatment for prostate cancer (PCa).Vesicourethral anastomosis (VUA) is a crucial step and either a conventional interrupted (IS) or a running (RS) suture is employed during radical prostatectomy (RP). Certainly, both RS and IS have advantages and limitations. The metanalysis revealed that potential advantages for RS compared to IS, especially for short-term outcomes such as catheterization time, extravasation rate, and anastomotic suture time. There were no significant differences for long-term outcomes (continence, incidence of vesicourethral anastomotic stenosis). Generally, the exciting evidence suggests that CS should be preferred over IS. However, this should be followed only if it is technically feasible and appropriate regarding the surgical approach. Both techniques seem to be safe and appropriate for the VUA, and the technique should be chosen based on individual experience and preference.

The investigators hypothesized that RS and IS may have different effects on voiding function and flow rate, even if they do not cause an anastomotic stenosis requiring intervention. Furthermore, there is no existing literature that compares RS and IS in terms of voiding function.This article focuses on one year uroflowmetric voiding parameters, urinary function (UF), and UF related bother function, urinary continence recovery as well as other secondary outcomes, including surgical parameters, perioperative morbidity and oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of clinically localised (pT1-pT2) prostate cancer
* must select the open radical prostatectomy procedure as a treatment option.

Exclusion Criteria:

* History of acute urinary retention
* History of urethral stricture

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Maximum flow rate (MFR) | preoperative and 1,3,6,12 months visits after surgery.
  Uroflowmetry is a noninvasive test that measures the rate of urine flow over time. Uroflowmetry involves a well-hydrated patient voiding into a uroflowmeter, which in turn generates a "flow curve." The flow curve enables the measurement of the MFR .A value of 15ml/sec or below is deemed to be outside the normal range.
Post-voiding residuel volume (PVR) | preoperative and 1,3,6,12 months visits after surgery.
  PVR is defined as the residual urine volume in the bladder following voiding, as calculated by ultrasound imaging. A volume of 150 cc or above is regarded as pathological.
Urinary function(UF) | preoperative and 1,3,6,12 months visits after surgery.
  Urinary function(UF) and urinary function-related bother: UF measured by the International Prostate Symptom Score [IPSS]) The IPSS is based on the answers to seven questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total score can therefore range from 0 to 35 . UF-related bother measured by the IPSS quality of life question with a response from 0 to 6.
Continence recovery | preoperative and 1,3,6,12 months visits after surgery.
  Urinary continence recovery defined as patient-reported use of zero pad or one security pad per day.

SECONDARY OUTCOMES:
Surgical parameters | During the operation
  Duration of vesico-urethral anastomosis time
Anastomotic extravasation | Postoperative day 5.
  Presence of anastomotic extravasation on first cystogram
Perioperative complications | Through study completion, an average of 1 year
  Clavien-Dindo scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Utku Can, Principal Investigator — Kartal Dr Lutfi Kirdar City Hospital
Locations (1):
- University of Health Sciences Kartal Dr. Lütfi Kırdar City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No